CLINICAL TRIAL: NCT00132379
Title: An Open-label, Phase I, Dose-escalation Study of ABR-217620 in Combination With Docetaxel in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: ABR-217620 in Combination With Docetaxel in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05762003
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — naptumomab estafenatox; CD3 Complex; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABR-217620; Drug: docetaxel

INTERVENTIONS:
Drug: ABR-217620 — 10.3, 16.5 or 22 mcg/kg, IV, daily 5 minute bolus injection for 4 consecutive day per cycle; up to 6 cycles
  Other Names: CD3; 5T4FabV18-SEA/E-120; naptumomab estafenatox; Anyara
Drug: docetaxel — 75mg/m^2, IV, single 60 minute infusion, beginning on Day 5 then every third week
  Other Names: Taxotere

SUMMARY:
The drug ABR-217620 is a combination of two proteins, one that recognizes tumor cells and one that triggers an attack on the tumor cells by activating some white blood cells belonging to the body's normal immune system. In animals, this results in an accumulation of white blood cells in the cancer that can fight the cancer. This study will test how much of the drug, in combination with docetaxel (an approved drug for treating non-small cell lung cancer [NSCLC]), can be given to patients with NSCLC without causing unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced NSCLC who have progressed on first line platin-based therapy or have failed on other treatment regimens or declined standard regimen.
* ECOG performance status 0 or 1.
* Adequate bone marrow function: absolute neutrophil count greater than or equal to 1500/mm3; WBC greater than or equal to 3000/mm3; platelets greater than or equal to 100,000/mm3; and hemoglobin greater than or equal to 10 g/dL.
* Adequate renal function: creatinine less than or equal to 1.5 x upper limit of normal (ULN).
* Adequate hepatic function: bilirubin less than ULN; and SGOT (AST) and SGPT (ALT) to less than 1.5 x ULN concomitant with alkaline phosphatase (ALP) less than 2.5 ULN.

Exclusion Criteria:

* Female patients who are pregnant or nursing or planning to become pregnant during the study. Fertile, sexually active women not willing to practice reliable contraception. Male patients with partners of childbearing potential not using acceptable contraceptive method.
* A serious uncontrolled medical disorder or active infection including unexplained fever (temperature greater than 100.5 degrees Fahrenheit or 38.1 degrees Celsius) that would impair the patient's ability to receive study treatment.
* Any concurrent malignancy, except for the following malignancies that may be included: non-melanoma skin cancer; cervical cancer in situ; ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) of breast; or past history of prostate cancer without clinical evidence of disease (includes patients receiving hormonal therapy).
* History of brain metastases, unless stable for more than 4 weeks, and not requiring steroid therapy and without clinical symptoms of brain metastases.
* Significant symptomatic cardiac disease including history (within past 6 months) or current unstable angina, congestive heart failure, or myocardial infarction; or patients with uncontrolled hypertension, or hypertension requiring treatment with more than 2 drugs.
* History of or current arrhythmias requiring treatment, except for non-specific, asymptomatic ST-T wave changes or extrasystoles.
* Seizure disorder requiring therapy.
* Treatment with beta-blockers, including topical therapy for glaucoma, during the 6-day treatment period (5-day treatment + 1 day in-patient follow-up), and within 5 days before start of ABR-217620 treatment.
* Simultaneous participation in any other investigational drug study or participation in a study less than 4 weeks before start of study treatment.
* Treatment with systemic or inhaled corticosteroids within 2 weeks before start of treatment.
* Treatment with anticoagulants, except when used to maintain the patency of a central venous line.
* Active autoimmune disease requiring therapy or any history of systemic lupus erythematosus or rheumatoid arthritis.
* Concurrent biological response modifiers (within 3 weeks of study entry) except for any type of erythropoetin.
* Chemo/radio/immunotherapy less than 4 weeks (6 weeks for mitomycin C and nitrosoureas) before start of treatment.
* Known allergy or hypersensitivity reactions to aminoglycosides (e.g., kanamycin).
* Known allergy or hypersensitivity reactions to docetaxel or other drugs formulated with polysorbate 80.
* Previous exposure to murine monoclonal antibody (with human anti-mouse antibody [HAMA] titer above detection limit at baseline) or known hypersensitivity to murine proteins.
* Major surgery within 3 weeks.
* Known history of HIV infection.
* Known chronic hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Side effect profile (based on blood pressure, body temperature, and laboratory tests) | Day 56 (Day 115 if undergo cycles 3/4)

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Days 1 and 4 of cycles 1 and 2
Immunological response | Day 56 (Day 115 if undergo cycles 3/4)
Changes in anti-SEA/E-120 levels | Day 56 (Day 115 if undergo cycles 3/4)
Objective response rate | Day 56 (Day 115 if undergo cycles 3/4)
Time to progression and Survival | Followed for up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Kilany, Study Director — Active Biotech AB
Locations (4):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States
- Onkologisk Klinik, Rigshospitalet, Copenhagen, Denmark
- Russia (2):
  - City Multifield Hospital #2, City Center of Intensive Pulmonology and Thoracic Surgery, Saint Petersburg
  - St. Petersburg Pavlov State Medical University, Saint Petersburg